CLINICAL TRIAL: NCT01910337
Title: Evaluation of Heart Rate Variability in Third Lower Molars Surgeries
Status: Completed | Type: Observational
Sponsor: Renata Martins da Silva Prado (Other)
Collaborators: University of Sao Paulo (Other)
Responsible Party: Sponsor-Investigator, Renata Martins da Silva Prado, 2926480, University of Sao Paulo
Organization: University of Sao Paulo (Other)
Other Study IDs: FR335167
Record Dates: First submitted 2013-07-25; First posted 2013-07-29 (Estimated); Last update posted 2013-07-29 (Estimated); Status verified 2013-07

CONDITIONS: Healthy Patients
Keywords: ASA I patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Screening: this first day, the patient will be evaluated with polar and blood pressure monitor. These data will be the basal one.
  Interventions: Device: Use the Polar Cardiac rate meter
- Intervation: One week later the screening, the patient underwent to the surgery to remove his lower third molar. In this day, will be analyzed 4 points: basal, after the anesthesia, after the avulsion and 20 minutes after the surgery.
  Interventions: Device: Use the Polar Cardiac rate meter
- Post operative: One week later the surgery, the patients will be evaluated again.
  Interventions: Device: Use the Polar Cardiac rate meter

INTERVENTIONS:
Device: Use the Polar Cardiac rate meter

SUMMARY:
The purpose of this study is to use heart rate variability as a monitor of cardiovascular safety during third molar surgeries, using the Polar heart rate-meter.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Patients (ASA I)
* Need to remove one of Lower Third Molar.

Exclusion Criteria:

* smoking
* pregnant

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 30 patients from the community sample in Dentistry School - University of Sao Paulo
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2011-06; Primary Completion 2011-11 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Evaluation of cardiac safety during third molar surgeries | 3 weekes

SECONDARY OUTCOMES:
study of heart rate variability during third molars surgeries with the Polar Cardiac Rate-meter. | 3 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Faculdade de Odontologia da Universidade de são Paulo, São Paulo, São Paulo, Brazil